CLINICAL TRIAL: NCT00758966
Title: A Proof-of-Concept, Multicenter, Randomized, Double-Blind, Parallel Study of Naltrexone Sustained-Release (SR) and/or Fluoxetine Therapy in the Treatment of Subjects With Obsessive-Compulsive Disorder (OCD)
Brief Title: Naltrexone SR and Fluoxetine Combination Therapy in Subjects With Obsessive-Compulsive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision- Financial Considerations
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NF-101
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD,; naltrexone,; fluoxetine,; obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluoxetine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NF (Naltrexone+Fluoxetine) (Experimental): Naltrexone SR 32 mg and fluoxetine 60 mg
  Interventions: Drug: Naltrexone 32 mg and fluoxetine 60 mg
- Fluoxetine (Active Comparator): Fluoxetine 60 mg
  Interventions: Drug: Fluoxetine 60 mg
- Naltrexone (Active Comparator): Naltrexone SR 32 mg
  Interventions: Drug: Naltrexone SR 32 mg

INTERVENTIONS:
Drug: Fluoxetine 60 mg — Two week titration followed by daily dosing of fluoxetine 60 mg for 8 weeks. Response is assessed at after 8 weeks. Responders will continue on fluoxetine 60 mg for an additional 6 weeks. Non-responders will have naltrexone SR 32 mg added to their therapy.
  Arms: Fluoxetine
Drug: Naltrexone 32 mg and fluoxetine 60 mg — Two week titration followed by daily dosing of naltrexone SR 32 mg and fluoxetine 60 mg for 8 weeks. Response is assessed at after 8 weeks. Responders will continue on a daily dose of naltrexone SR 32 mg and fluoxetine 60 mg for an additional 6 weeks. Non-responders will have their daily dose adjusted to naltrexone SR 48 mg and fluoxetine 80 mg.
  Arms: NF (Naltrexone+Fluoxetine)
Drug: Naltrexone SR 32 mg — Two week titration followed by daily dosing of naltrexone SR 32 mg for 8 weeks. Response is assessed at after 8 weeks. Responders will continue on naltrexone SR 32 mg for an additional 6 weeks. Non-responders will have fluoxetine 60 mg added to their therapy.
  Arms: Naltrexone

SUMMARY:
The purpose of this study is to determine if the combination of naltrexone SR and fluoxetine is more effective in treating the symptoms of obsessive-compulsive disorder (OCD)than either fluoxetine alone or naltrexone SR alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 60 years of age (inclusive)
* Outpatients with a current diagnosis of OCD that have received previous therapy
* Negative serum pregnancy test as screening in women of child-bearing potential
* If a woman of child-bearing potential, must agreed to use an acceptable and effective form of contraception
* No clinically significant abnormality on electrocardiogram (ECG)
* No clinically significant laboratory abnormality at screening
* Negative urine drug screen
* Must be considered reliable and possess a level of understanding that enables the subject to provide written informed consent and to comply with protocol procedures and schedule

Exclusion Criteria:

* Diagnosis of substance dependence
* Diagnosis of substance abuse (except for nicotine and caffeine)
* Serious or unstable medical illnesses
* Lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, anorexia nervosa, Pervasive Developmental Disorder (PDD), Asperger's Syndrome or the presence of antisocial or borderline personality disorder
* Diagnosis of tic disorder or Tourette's Syndrome
* Subjects diagnosed with impulse control disorder
* Known sensitivity or allergic reaction to either naltrexone or fluoxetine
* Any condition which in the opinion of the investigator or Sponsor makes the subject unsuitable for inclusion in the study
* Immediate family of investigators, study personnel or Sponsor representatives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the mean change from baseline to Week 10 in total Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score between the combination treatment group versus fluoxetine alone and naltrexone SR alone | Baseline to Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Apter, MD, PA, Principal Investigator — Global Medical Institutes, LLC; Ward Smith, MD, Principal Investigator — Summit Research Network, Inc.; Vishaal Mehra, MD, Principal Investigator — California Clinical Trials; Naresh P Emmanuel, MD, Principal Investigator — Carolina Clinical Research Services; Mohammad Bari, MD, Principal Investigator — Synergy Clinical Research; Robert Riesenberg, MD, Principal Investigator — Atlanta Center for Medical Research; Teresa Pigott, MD, Principal Investigator — University of Florida, Dept Of Psychiatry; Andrew W Goddard, MD, Principal Investigator — Indiana University School of Medicine; Al Rivera, MD, Principal Investigator — Community Research; Jeffrey S Simon, MD, Principal Investigator — Northbrooke Research Center; Zinoviy Benzar, MD, Principal Investigator — Brooklyn Medical Institute
Locations (11):
- United States (11):
  - Synergy Clinical Research, National City, California
  - California Clinical Trials, San Diego, California
  - University of Florida, Department of Psychiatry, Gainesville, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Global Medical Institute, LLC, Princeton, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Community Research, Cincinnati, Ohio
  - Summit Research Network, Inc., Portland, Oregon
  - Carolina Clinical Research Services, Columbia, South Carolina
  - Northbrooke Research Center, Brown Deer, Wisconsin